CLINICAL TRIAL: NCT00131859
Title: Diffusion-Tensor Magnetic Resonance Imaging and the Evaluation of Perinatal Brain Injury
Brief Title: Diffusion-Tensor Magnetic Resonance Imaging (MRI) and the Evaluation of Perinatal Brain Injury
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Ernie Graham, M.D., Johns Hopkins University School of Medicine
Other Study IDs: 04-08-31-01
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Brain Injury, Fetus and Neonate
Keywords: Perinatal brain injury; Diffusion-tensor imaging
MeSH Terms: conditions — Brain Injuries | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Diffusion-tensor imaging — Obtain a Diffusion tensor MRI of brain.
  Other Names: No other names applicable.

SUMMARY:
The researchers' objective is to use diffusion-tensor imaging (DTI) to evaluate infants diagnosed with cerebral white matter injury during the neonatal period and identify antenatal risk factors, electronic fetal heart rate monitoring abnormalities, and umbilical arterial gas results that are associated with cerebral white matter injury. The researchers' hypothesis is that this new imaging technique will help us better understand how these devastating injuries occur.

DETAILED DESCRIPTION:
Maternal and neonatal data will be collected as well as the umbilical arterial gas results and the electronic fetal heart rate tracing of the labor. Infants will have a head ultrasound at 24-72 hours, 10-14 days, and at 4-6 weeks to look for cerebral white matter injury, as standard of care. All infants with a birth weight < 1500 grams will be offered DTI, and infants > 1500 grams with white matter injury diagnosed by ultrasound will be imaged as well as the subsequent delivery born within 7 days of that gestational age without brain injury. All infants will have the DTI brain scan at 12-18 months of age corrected for the degree of prematurity, and will also have a formal neurological assessment at that time.

ELIGIBILITY:
Inclusion Criteria:

* All infants born at our hospital at < 1500 grams
* All infants born at our hospital at > 1500 grams with brain injury or severe metabolic acidosis

Exclusion Criteria:

* Major congenital malformations
* Chromosomal abnormality

Ages: 23 Weeks to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates < 1500 grams, with suspected brain injury, and with severe metabolic acidosis
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2004-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Diffusion-tensor imaging differences between brain injured cases and controls without brain injury | 2 years

SECONDARY OUTCOMES:
Umbilical cord gas results | 2 years
Placental pathology | 2 years
Electronic fetal monitoring | 2 years
Nucleated red blood cells | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ernest M Graham, M.D., Principal Investigator — Johns Hopkins Univ; Dept. of Gyn-Ob
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States